CLINICAL TRIAL: NCT06428721
Title: The Preventive Role of Fractionated Laser Resurfacing Against Actinic Neoplasia in an At-Risk Geriatric Population
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Wright State University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2023-346
Record Dates: First submitted 2024-05-20; First posted 2024-05-24 (Actual); Last update posted 2024-07-24 (Actual); Status verified 2024-07

CONDITIONS: Actinic Keratoses; Aging; Non-Melanoma Skin Cancer
MeSH Terms: conditions — Keratosis, Actinic

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Fractionated Laser Resurfacing - Right Arm (Experimental): Right forearm treatment of fractionated laser resurfacing.
  Interventions: Device: Fractionated Laser Resurfacing
- Fractionated Laser Resurfacing - Left Arm (Experimental): Left forearm treatment of fractionated laser resurfacing.
  Interventions: Device: Fractionated Laser Resurfacing

INTERVENTIONS:
Device: Fractionated Laser Resurfacing — A rejuvenating laser that makes tiny holes in the very superficial part of the skin.

SUMMARY:
The purpose of this study is to determine if the Fractionated Laser Resurfacing (FLR) procedure can protect one forearm/wrist from precancerous actinic keratosis (AKs) as well as prevent skin cancer in older subjects with active AKs. This study builds on a similar study ongoing at the Dayton Veterans Administration dermatology clinic. This study is also testing if a photograph of the skin can be used to predict where the AKs and an skin cancers will form.

ELIGIBILITY:
Inclusion Criteria:

* Adult Males and Females aged 60 and older
* Have at least 5 AKs on each forearm/wrist, but no more than 10 to allow for easy monitoring
* Skin type fair (Fitzpatrick I-II)
* Females must be post-menopausal and not be on systemic hormone replacement therapy
* Able to comprehend procedures and risks

Exclusion Criteria:

* More than 10 AKs on an extremity
* AKs that are large (2-3+, hyperkeratotic grade 3 lesions)
* AKs that are very thick (>3 mm)
* Medical history of diabetes
* History of poor wound healing or scarring
* Large tattoos that can interfere with study
* Other serious health issues and other skin diseases that could interfere with the study
* Recent (within 1 year) field therapies such as efudex cream or PDT to forearms/wrists.
* Planning to leave region in next 5 years
* Subjects with allergies to xylocaine will be excluded if they need this topical anesthetic.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-03-20 (Actual); Primary Completion 2031-12 (Estimated); Study Completion 2031-12 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in the number of actinic keratosis due to FLR treatment. | Up to 5 years
  Investigator will assess the number of actinic keratosis on both forearms at each visit.
Change from baseline in the number of non-melanoma skin cancers due to FLR treatment. | Up to 5 years
  Investigator will assess the number of actinic keratosis on both forearms at each visit.

SECONDARY OUTCOMES:
Skin dysplasia change, in regards to actinic keratosis, from baseline due to FLR treatment. | Up to 5 years
  Investigator will use the scattering patterns of light to assess the number of actinic keratosis on both forearms at each visit.
Skin dysplasia change, in regards to non-melanoma skin cancer, from baseline due to FLR treatment. | Up to 5 years
  Investigator will use the scattering patterns of light to assess the number of actinic keratosis on both forearms at each visit.

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Travers, MD, PhD, Principal Investigator — Wright State University
Locations (1):
- Wright State Physicians, Fairborn, Ohio, United States